CLINICAL TRIAL: NCT02131467
Title: An Open-label Phase 2a Study to Evaluate the Safety and Tolerability of Perampanel (E2007) in Subjects With Cervical Dystonia (SAFE-Per CD)
Brief Title: Safety and Tolerability of Perampanel in Cervical Dystonia
Acronym: SAFE-PER-CD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Dystonia Study Group (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-5864.4
Record Dates: First submitted 2014-04-23; First posted 2014-05-06 (Estimated); Last update posted 2020-04-07 (Actual); Status verified 2020-04

CONDITIONS: Cervical Dystonia
MeSH Terms: conditions — Torticollis | interventions — perampanel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Perampanel (Experimental): Perampanel 2 mg tablets will be initiated once daily at bedtime. The dose will be titrated over 6 weeks starting at 2 mg OD at baseline visit for 1 week, followed by 2mg increases every 1 week to a maximum of 12 mg/day. If side effects occur then patients will be decreased to previous dose level. If unable to tolerate increases, patients will enter the maintenance phase at previously tolerated dose, for minimum 4 weeks. Patients reaching 12 mg (maximal dose) will be maintained at that dose for 4 weeks. Taper will be over 2 weeks 1 tablet every 2 days from a maximum of 6 tablets per day to stop.
  Interventions: Drug: Perampanel

INTERVENTIONS:
Drug: Perampanel — oral drug

SUMMARY:
Cervical dystonia (CD) is the most common focal dystonia. Currently there are no effective oral medications for the treatment of CD. While botulinum toxin injections improve symptoms, they require repeated injections by a trained physician and some patients stop responding to injections or never respond at all. Therefore, alternative treatment options for CD are needed. One new agent is a drug that targets glutamate receptors that are thought to be involved dystonia. This drug, perampanel, was originally developed for epilepsy and is licensed for use in the USA and Canada for treating epilepsy. The purpose of this study is to test the effectiveness of perampanel in treating the symptoms of CD.

DETAILED DESCRIPTION:
Idiopathic cervical dystonia (CD) is the most common form of focal dystonia with a prevalence of approximately 60 cases per million population.(Nutt et al.,1988). Current oral medical treatments for CD have variable efficacy and often with marked side effects. Botulinum toxin injections may be more effective than pharmacological therapies, and are currently the best available therapeutic option. However, repeat injections, administered by a physician trained in this area are required every 3-4 months.(Brans et al.,1996) This can often be difficult and costly for patients. Furthermore, there are subgroups of patients who simply do not respond to this treatment and between 5-20% of patients may become secondary non responders due to the development of blocking antibodies to the botulinum toxin.(Mejia et al., 2005) Thus, new therapeutic options are required.

The neural mechanisms underlying idiopathic dystonia are not well known. Classical basal ganglia circuitry models predict underactivity of the output regions of the basal ganglia, the medial globus pallidus and substantia nigra pars reticulata (;Mitchell et al 1990). In subjects with dystonia undergoing DBS, intraoperative recordings have demonstrated underactivity of the medial globus pallidus (Vitek et al, 1999, Lozano et al 1997). One mechanism responsible for these basal ganglia output changes may be overactivity of corticostriatal glutamatergic pathways, as similar neural mechanism are thought to underlie other hyperkinetic movements (Brotchie 2005). The best studied hyperkinetic movement disorder is levodopa-induced dyskinesia in Parkinson's disease in which dystonia, often of the head and neck, may occur. In animal models of levodopa-induced dyskinesia, increased striatal glutamatergic signaling via alpha-amino-2,3-dihydro-5-methyl-3-oxo-4-isoxazolepropanoic acid (AMPA) receptors has been demonstrated (Perier et al 2002, Silverdale et al 2010). To date there are few validated animal models of idiopathic dystonia. However, one model that has been use for pharmacological studies, and the results extrapolated to idiopathic dystonia, is the paroxysmal dt(sz) dystonic hamster (Loscher and Richter 1998). In this model, intrastriatal and systemic injection of NBQX a selective AMPA receptor antagonist reduced dystonic severity (Richter et al 1993, Sander and Richter 2002, Kohling et al 2004). Other studies have suggested that cerebellar outflow pathways, using AMPA receptors may also mediate dystonic symptoms. Thus the excitatory amino-acid kainite injected into rodent cerebellar vermis resulted in dystonic symptoms, an effect revered by NBQX, suggesting an action on AMPA receptors (Pizoli et al 2002). Thus AMPA receptor antagonists may alleviate dystonia.

To date, clinical studies using glutamate antagonists in CD have been limited due to lack of available drugs. A single 6-week open-label pilot study of the non-selective glutamate antagonist riluzole (50 mg twice a day) in six patients with cervical dystonia (CD) reported a 26% improvement in CD with no side-effects (Muller et al 2002).

The aim of this study is to conduct a multicentre phase I/IIa open label study to determine the safety and tolerability of the AMPA antagonist, perampanel in subjects with primary cervical dystonia. Exploratory analysis will determine effects on dystonia disability and subjective measures including quality of life and global impression of change. The importance of such an initial safety study is due to the lack of knowledge related to the use of this class of drug (AMPA antagonist) in this population of patients. The longer term aim is thus to generate preliminary data for further randomised controlled efficacy studies.

ELIGIBILITY:
Inclusion Criteria:

* • 18-65 year old male and female patients with primary cervical dystonia.

  * Subject may be untreated with botulinum toxin; treated with botulinum toxin but who are at least 8 weeks (+ 1 week) from a previous injection; or who have experienced an insufficient response to botulinum toxin in the opinion of the enrolling investigator. Note: We will aim to include subjects who have a stable response that lasts 12 weeks or longer.
  * Subjects may be on stable anti-dystonia treatment (for at least one month) including anticholinergics, baclofen, and anxiolytics including benzodiazepines.

Exclusion Criteria:

* Secondary cervical dystonia,

  * Significant dystonia in body areas other than cervical region,
  * Cognitive impairment (e.g., Montreal Cognitive assessment (MOCA) < 26);
  * Active psychosis;
  * History of aggression;
  * Active depression (Hamilton Depression Rating Scale (HDRS) score ≥ 12).
  * Current abuse of alcohol or subjects who do not agree to avoid alcohol during treatment,
  * Substance abuse (current or prior);
  * Active infection,
  * Hypersensitivity to perampanel,
  * Significant renal dysfunction (Creatinine clearance < 50ml/min),
  * Significant laboratory abnormalities (ALT or AST greater than twice normal value; elevated bilirubin, active liver disease: hepatitis, cholestasis, cirrhosis, etc.),
  * Significant medical illness,
  * Women who are pregnant or plan to become pregnant, women who are breastfeeding,
  * Subjects who do not agree to avoid consumption of grapefruit or grapefruit-containing products throughout the study,
  * Galactose intolerance, the Lapp lactase deficiency or glucose-galactose malabsorption
  * Use of prohibited medications known to be inducers of CYP3A including, but not limited to: rifampicin, troglitazone, St John's Wort, efavirenz, nevirapine, barbiturates, glucocorticoids (other than topical usage), modafinil, pioglitazone, and rifabutin; and any other interactions as per Product Monograph

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2017-09-01 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Number of subjects able to remain on study drug for minimum of 4 weeks. | Measured at week 12.
  Tolerability will be assessed by counting number of subjects able to remain on drug

SECONDARY OUTCOMES:
Safety will be evaluated as the cumulative number of new adverse events collected at each visit from Baseline to visit 4 | Adverse events at study visits weeks 0, 2, 6, 8, 9, 10 and 12
  Adverse events will be assessed at each visit by direct questioning patients, measuring weight, vital signs, Hamilton depression scale and laboratory tests and ECG

OTHER OUTCOMES:
Change from baseline to end of maintenance in Toronto Western Spasmodic Torticollis Rating Scale (TWSTRS) | week 12
  The TWSTRS is a validated rating scale that measures disability due to cervical dystonia.
CDIP58 | week 12
  Change in impact of Cervical Dystonia on quality of life using the CDIP 58 from baseline to end of maintenance
CGI | week 12
  Change in Clinical global Impression (CGI) of Cervical Dystonia severity (patient and investigator) from baseline to end of maintenance

CONTACTS AND LOCATIONS:
Overall Officials: Susan H Fox, MRCP(UK), PhD, Principal Investigator — University Health Network, Toronto
Locations (5):
- United States (4):
  - Emory University School of Medicine, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - Beth Israel Medical Center, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
- Toronto Western Hospital, Toronto, Ontario, Canada